CLINICAL TRIAL: NCT01926015
Title: Post-marketing, Randomized, Open-label Study to Assess the Immunogenicity and Safety of Concomitant Administration of V260 and Diphtheria, Tetanus, Pertussis and Inactivated Poliovirus Vaccine (DTP-IPV) in Japanese Healthy Infants
Brief Title: Immunogenicity and Safety of Concomitant Administration of RotaTeq™ (V260) and the Diphtheria, Tetanus, Pertussis and Inactivated Poliovirus Vaccine (DTP-IPV) in Healthy Japanese Infants (V260-060)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V260-060; 132252 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2013-08-16; First posted 2013-08-20 (Estimated); Results first posted 2015-04-09 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-10

CONDITIONS: Rotavirus Disease
MeSH Terms: conditions — Rotavirus Infections | interventions — RotaTeq; Rotavirus Vaccines; DTP-IPV-Hib vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Concomitant RotaTeq™ and DTP-IPV (Experimental): RotaTeq™ (2 mL oral dose) and DTP-IPV (0.5 mL subcutaneous injection) administered concomitantly at Visit 2 (>=4 weeks after Visit 1), Visit 4 (6-8 weeks after Visit 2), and Visit 6 (6-8 weeks after Visit 4).
  Interventions: Biological: RotaTeq™ (V260); Biological: DTP-IPV
- Staggered RotaTeq™ and DTP-IPV (Active Comparator): RotaTeq™ (2 mL oral dose) administered at Visit 1 (Day 1), Visit 3 (6-8 weeks after Visit 1), and Visit 5 (6-8 weeks after Visit 3) and DTP-IPV (0.5 mL subcutaneous injection) administered at Visit 2 (>=4 weeks after Visit 1), Visit 4 (6-8 weeks after Visit 2), and Visit 6 (6-8 weeks after Visit 4).
  Interventions: Biological: RotaTeq™ (V260); Biological: DTP-IPV

INTERVENTIONS:
Biological: RotaTeq™ (V260) — Live, oral, pentavalent vaccine containing 5 human-bovine reassortant rotavirus strains
  Other Names: RotaTeq™
Biological: DTP-IPV — Diphtheria, tetanus, pertussis, inactivated polio vaccine used as part of the Japanese vaccination schedule
  Other Names: Tetrabik™; BIKEN

SUMMARY:
The study will evaluate the immunogenicity of the Diphtheria, Tetanus, Pertussis and Inactivated Poliovirus Vaccine (DTP-IPV) with concomitant administration of RotaTeq™ (V260) in healthy Japanese infants. The hypothesis to be tested is that the antibody response rates to DTP-IPV with concomitant administration of RotaTeq™ are non-inferior to those with staggered administration of RotaTeq™.

ELIGIBILITY:
Inclusion Criteria:

* Japanese participant
* Age 6 weeks through <11 weeks (42 to 76 days from date of birth) at Visit 1

Exclusion Criteria:

* History of hypersensitivity and/or anaphylaxis to any of the product ingredients in V260 or DTP-IPV
* Gastrointestinal disorder, growth retardation, or failure to thrive
* History of intussusception
* Untreated congenital gastrointestinal disorder (such as Meckel diverticulum)
* Known or suspected impairment of immunological function, including severe immunodeficiency (SCID)
* Cardiovascular, renal, liver, or blood disease
* History of convulsion
* Undergoing immunosuppressive therapy or living with a close relative with congenital immune deficiency
* Prior vaccination with rotavirus vaccine and/or DTP-IPV vaccine
* Live vaccine received within 28 days or inactivated vaccine received within 7 days
* At high risk for tuberculosis exposure

Ages: 6 Weeks to 11 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 192 (Actual)
Dates: Start 2013-09-19 (Actual); Primary Completion 2014-06-06 (Actual); Study Completion 2014-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Tanaka Y, Yokokawa R, Rong HS, Kishino H, Stek JE, Nelson M, Lawrence J. Concomitant administration of diphtheria, tetanus, acellular pertussis and inactivated poliovirus vaccine derived from Sabin strains (DTaP-sIPV) with pentavalent rotavirus vaccine in Japanese infants. Hum Vaccin Immunother. 2017 Jun 3;13(6):1-7. doi: 10.1080/21645515.2017.1279769. Epub 2017 Jan 31. PMID 28140752
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=V260-060&kw=V260-060&tab=access

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Concomitant RotaTeq™ and DTP-IPV | Staggered RotaTeq™ and DTP-IPV
Started | 96 (Participants who passed all entry criteria and who were randomized into the study) | 96 (Participants who passed all entry criteria and who were randomized into the study)
Received >=1 Vaccination | 94 | 96
Completed | 94 | 95
Not Completed | 2 | 1
Not completed — Withdrawal by parent/guardian | 0 | 1
Not completed — Randomized not treated | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Concomitant RotaTeq™ and DTP-IPV | Staggered RotaTeq™ and DTP-IPV | Total
Number analyzed (Participants) | 96 | 96 | 192
Age, Continuous [Median (Full Range); unit: Weeks] | 8 [6 to 10] | 9 [6 to 10] | 9 [6 to 10]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 41 | 88
  Male | 49 | 55 | 104

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Seroresponse for Diphtheria Toxin, Tetanus Toxin, Pertussis Filamentous Hemagglutinin (FHA), and Poliovirus Type 1, 2, and 3
Description: Participant serum was collected for determination of antibody responses. Threshold levels for seroresponse were the following: Diphtheria Toxin, >=0.1 International Units (IU)/mL; Tetanus Toxin, >=0.01 IU/mL; Pertussis Toxin and Pertussis FHA, >=10 Enzyme Units (EU)/mL; Poliovirus Types 1, 2, and 3, neutralizing antibody (NA) titer >=8.
Time Frame: 4 to 6 weeks after the third dose of DTP-IPV
Population: The per-protocol population included participants who received the 3 scheduled doses of DTP-IPV according to guidelines and did not have an important protocol deviation that may substantially affect the results of the endpoint
Measure: Number; unit: Percentage of participants
Arm/Group | Concomitant RotaTeq™ and DTP-IPV | Staggered RotaTeq™ and DTP-IPV
Number analyzed (Participants) | 93 | 94
Percentage of participants
  Diphtheria Toxin >=0.1 IU/mL | 100 | 100
  Tetanus Toxin >=0.01 IU/mL | 100 | 100
  Pertussis Toxin >=10 EU/mL | 100 | 100
  Pertussis FHA >=10 EU/mL | 100 | 100
  Poliovirus Type 1 NA >=8 | 100 | 100
  Poliovirus Type 2 NA >=8 | 100 | 100
  Poliovirus Type 3 NA >=8 | 100 | 100
Statistical Analysis 1: Comparison: Concomitant RotaTeq™ and DTP-IPV vs Staggered RotaTeq™ and DTP-IPV; Diphtheria Toxin >=0.1 IU/mL; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower bound of the 95% confidence interval of the percentage difference, excluding a difference >=10%, is >=-0.10; p < 0.001, Miettinen and Nurminen; Difference in percentage = 0.0, 95% CI 2-sided [-3.99 to 3.95]
Statistical Analysis 2: Comparison: Concomitant RotaTeq™ and DTP-IPV vs Staggered RotaTeq™ and DTP-IPV; Tetanus Toxin >=0.01 IU/mL; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in percentage = 0.0, 95% CI 2-sided [-3.99 to 3.95]
Statistical Analysis 3: Comparison: Concomitant RotaTeq™ and DTP-IPV vs Staggered RotaTeq™ and DTP-IPV; Pertussis Toxin >=10 EU/mL; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in percentage = 0.0, 95% CI 2-sided [-3.99 to 3.95]
Statistical Analysis 4: Comparison: Concomitant RotaTeq™ and DTP-IPV vs Staggered RotaTeq™ and DTP-IPV; Pertussis FHA >=10 EU/mL; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in percentage = 0.0, 95% CI 2-sided [-3.99 to 3.95]
Statistical Analysis 5: Comparison: Concomitant RotaTeq™ and DTP-IPV vs Staggered RotaTeq™ and DTP-IPV; Poliovirus Type 1 NA >=8; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in percentage = 0.0, 95% CI 2-sided [-3.99 to 3.95]
Statistical Analysis 6: Comparison: Concomitant RotaTeq™ and DTP-IPV vs Staggered RotaTeq™ and DTP-IPV; Poliovirus Type 2 NA >=8; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in percentage = 0.0, 95% CI 2-sided [-3.99 to 3.95]
Statistical Analysis 7: Comparison: Concomitant RotaTeq™ and DTP-IPV vs Staggered RotaTeq™ and DTP-IPV; Poliovirus Type 3 NA >=8; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in percentage = 0.0, 95% CI 2-sided [-3.99 to 3.95]

2. Secondary Outcome: Percentage of Participants Reporting an Adverse Event With Incidence >=1%
Description: An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation subject administered study drug and which does not necessarily have to have a causal relationship with this treatment. Any worsening of a preexisting condition that is temporally associated with the use of the study drug is also an adverse event. Adverse events with an incidence >=1% in either treatment group were recorded.
Time Frame: Up to 14 days after any of the 6 study visits
Population: The safety population included randomized participants who received >=1 dose of study vaccine and had safety follow-up. Each participant was were counted only once overall.
Measure: Number; unit: Percentage of participants
Arm/Group | Concomitant RotaTeq™ and DTP-IPV | Staggered RotaTeq™ and DTP-IPV
Number analyzed (Participants) | 94 | 96
Percentage of participants | 68.1 | 86.5

3. Secondary Outcome: Percentage of Participants Reporting an Adverse Event of Special Interest: Fever
Description: An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation subject administered study drug and which does not necessarily have to have a causal relationship with this treatment. Any worsening of a preexisting condition that is temporally associated with the use of the study drug is also an adverse event. Adverse events of special interest included fever, diarrhea, vomiting, and injection-site adverse events.
Time Frame: Period 1 (up to 14 days after Visit 1 [V1] or V2), Period 2 (up to 14 days after V3 or V4), Period 3 (up to 14 days after V5 or V6), and Overall (up to 14 days after any visit)
Population: The safety population included randomized participants who received >=1 dose of study vaccine and had safety follow-up. Each participant was counted only once within a study Period and only once Overall.
Measure: Number; unit: Percentage of participants
Arm/Group | Concomitant RotaTeq™ and DTP-IPV | Staggered RotaTeq™ and DTP-IPV
Number analyzed (Participants) | 94 | 96
Percentage of participants
  Period 1 (up to 14 days after V1 or V2) (n=94, 96) | 5.3 | 6.3
  Period 2 (up to 14 days after V3 or V4) (n=94, 96) | 1.1 | 12.5
  Period 3 (up to 14 days after V5 or V6)(n=94, 95) | 4.3 | 6.3
  Overall (up to 14 days after any visit)(n=94, 96) | 10.6 | 22.9

4. Secondary Outcome: Percentage of Participants Reporting an Adverse Event of Special Interest: Diarrhea
Description: as for outcome 3
Time Frame: as for outcome 3
Population: The safety population included randomized participants who received >=1 dose of study vaccine and had safety follow-up. Participants are counted only once within a study Period and only once Overall.
Measure: Number; unit: Percentage of participants
Arm/Group | Concomitant RotaTeq™ and DTP-IPV | Staggered RotaTeq™ and DTP-IPV
Number analyzed (Participants) | 94 | 96
Percentage of participants
  Period 1 (up to 14 days after V1 or V2) (n=94, 96) | 17.0 | 31.3
  Period 2 (up to 14 days after V3 or V4) (n=94, 96) | 10.6 | 20.8
  Period 3 (up to 14 days after V5 or V6) (n=94, 95) | 7.4 | 18.9
  Overall (up to 14 days after any visit)(n=94, 96) | 25.5 | 46.9

5. Secondary Outcome: Percentage of Participants Reporting an Adverse Event of Special Interest: Vomiting
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Concomitant RotaTeq™ and DTP-IPV | Staggered RotaTeq™ and DTP-IPV
Number analyzed (Participants) | 94 | 96
Percentage of participants
  Period 1 (up to 14 days after V1 or V2) (n=94, 96) | 5.3 | 9.4
  Period 2 (up to 14 days after V3 or V4) (n=94, 96) | 3.2 | 6.3
  Period 3 (up to 14 days after V5 or V6) (n=94, 95) | 1.1 | 4.2
  Overall (up to 14 days after any visit) (n=94, 96) | 8.5 | 16.7

6. Secondary Outcome: Percentage of Participants Reporting an Adverse Event of Special Interest: Injection-site Adverse Events
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Concomitant RotaTeq™ and DTP-IPV | Staggered RotaTeq™ and DTP-IPV
Number analyzed (Participants) | 94 | 96
Percentage of participants
  Period 1 (up to 14 days after V1 or V2) (n=94, 96) | 2.1 | 4.2
  Period 2 (up to 14 days after V3 or V4) (n=94, 96) | 0.0 | 8.3
  Period 3 (up to 14 days after V5 or V6) (n=94, 95) | 0.0 | 2.1
  Overall (up to 14 days after any visit) (n=94, 96) | 2.1 | 10.4

7. Secondary Outcome: Geometric Mean Titers for Diphtheria Toxin Antibody
Description: Participant serum was collected for determination of antibody responses before the first dose of study vaccine (Baseline) and 4 to 6 weeks after the third dose of DTP-IPV
Time Frame: Predose (Baseline) and 4 to 6 weeks after the third dose of DTP-IPV
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Concomitant RotaTeq™ and DTP-IPV | Staggered RotaTeq™ and DTP-IPV
Number analyzed (Participants) | 93 | 94
IU/mL
  Baseline | 0.025 [0.018 to 0.034] | 0.019 [0.014 to 0.026]
  4 to 6 weeks after the third dose of DTP-IPV | 2.377 [2.032 to 2.780] | 2.493 [2.165 to 2.871]

8. Secondary Outcome: Geometric Mean Titers for Tetanus Toxin Antibody
Description: as for outcome 7
Time Frame: Predose (Baseline) and 4 to 6 weeks after the third dose of DTP-IPV
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Concomitant RotaTeq™ and DTP-IPV | Staggered RotaTeq™ and DTP-IPV
Number analyzed (Participants) | 93 | 94
IU/mL
  Baseline | 0.082 [0.059 to 0.114] | 0.093 [0.067 to 0.128]
  4 to 6 weeks after the third dose of DTP-IPV | 1.001 [0.702 to 1.428] | 1.338 [1.009 to 1.774]

9. Secondary Outcome: Geometric Mean Titers for Pertussis Toxin Antibody
Description: as for outcome 7
Time Frame: Predose (Baseline) and 4 to 6 weeks after the third dose of DTP-IPV
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Concomitant RotaTeq™ and DTP-IPV | Staggered RotaTeq™ and DTP-IPV
Number analyzed (Participants) | 93 | 94
EU/mL
  Baseline | 2.670 [2.143 to 3.328] | 2.757 [2.278 to 3.338]
  4 to 6 weeks after the third dose of DTP-IPV | 198.811 [177.430 to 222.768] | 241.857 [218.225 to 268.049]

10. Secondary Outcome: Geometric Mean Titers for Pertussis FHA Antibody
Description: as for outcome 7
Time Frame: Predose (Baseline) and 4 to 6 weeks after the third dose of DTP-IPV
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Concomitant RotaTeq™ and DTP-IPV | Staggered RotaTeq™ and DTP-IPV
Number analyzed (Participants) | 93 | 94
EU/mL
  Baseline | 7.513 [6.285 to 8.980] | 6.951 [5.703 to 8.472]
  4 to 6 weeks after the third dose of DTP-IPV | 77.386 [67.959 to 88.119] | 88.275 [76.065 to 102.445]

11. Secondary Outcome: Geometric Mean Titers for Poliovirus Type 1 Antibody
Description: Participant serum was collected for determination of antibody responses before the first dose of study vaccine (Baseline) and 4 to 6 weeks after the third dose of DTP-IPV. Poliovirus antibodies are expressed as neutralizing antibody (NA) titers.
Time Frame: Predose (Baseline) and 4 to 6 weeks after the third dose of DTP-IPV
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: NA Titer
Arm/Group | Concomitant RotaTeq™ and DTP-IPV | Staggered RotaTeq™ and DTP-IPV
Number analyzed (Participants) | 93 | 94
NA Titer
  Baseline | 23.5 [17.21 to 32.05] | 21.1 [15.47 to 28.76]
  4 to 6 weeks after the third dose of DTP-IPV | 1578 [1237.3 to 2012.0] | 1703 [1314.4 to 2207.0]

12. Secondary Outcome: Geometric Mean Titers for Poliovirus Type 2 Antibody
Description: as for outcome 11
Time Frame: Predose (Baseline) and 4 to 6 weeks after the third dose of DTP-IPV
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: NA Titer
Arm/Group | Concomitant RotaTeq™ and DTP-IPV | Staggered RotaTeq™ and DTP-IPV
Number analyzed (Participants) | 93 | 94
NA Titer
  Baseline | 32.0 [23.97 to 42.72] | 27.8 [20.64 to 37.49]
  4 to 6 weeks after the third dose of DTP-IPV | 2886 [2346.9 to 3547.8] | 3259 [2678.2 to 3965.8]

13. Secondary Outcome: Geometric Mean Titers for Poliovirus Type 3 Antibody
Description: as for outcome 11
Time Frame: Predose (Baseline) and 4 to 6 weeks after the third dose of DTP-IPV
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: NA Titer
Arm/Group | Concomitant RotaTeq™ and DTP-IPV | Staggered RotaTeq™ and DTP-IPV
Number analyzed (Participants) | 93 | 94
NA Titer
  Baseline | 3.9 [3.43 to 4.43] | 4.8 [3.92 to 5.85]
  4 to 6 weeks after the third dose of DTP-IPV | 2377 [1973.1 to 2864.0] | 2671 [2193.5 to 3251.5]

ADVERSE EVENTS:
Time Frame: All adverse events: up to 14 days after any study visit; all deaths, vaccine-related serious adverse events, overdoses, and intussusception: up to 26 weeks after Visit 1
Description: The safety population included randomized participants who received >=1 dose of study vaccine and had safety follow-up
Arm/Group | Concomitant RotaTeq™ and DTP-IPV | Staggered RotaTeq™ and DTP-IPV
Serious Adverse Events (participants affected / at risk) | 0/94 | 2/96
Other Adverse Events (participants affected / at risk) | 57/94 | 79/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Concomitant RotaTeq™ and DTP-IPV (N=94) | Staggered RotaTeq™ and DTP-IPV (N=96)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Concomitant RotaTeq™ and DTP-IPV (N=94) | Staggered RotaTeq™ and DTP-IPV (N=96)
Diarrhoea (Gastrointestinal disorders) | 24 | 45
Infantile spitting up (Gastrointestinal disorders) | 0 | 6
Vomiting (Gastrointestinal disorders) | 8 | 16
Injection site erythema (General disorders) | 2 | 5
Pyrexia (General disorders) | 10 | 22
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 9 | 12
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 6 | 9
Eczema infantile (Skin and subcutaneous tissue disorders) | 7 | 7
Bronchitis (Infections and infestations) | 5 | 4
Conjunctivitis (Infections and infestations) | 2 | 6
Nasopharyngitis (Infections and infestations) | 7 | 20
Upper respiratory tract infection (Infections and infestations) | 9 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.